CLINICAL TRIAL: NCT05562141
Title: Oxidative Stress in the Patient With Peroperative Analgesia by Intravenous Lidocaine
Acronym: OSPAIL
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR220194-OSPAIL
Record Dates: First submitted 2022-09-23; First posted 2022-09-30 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Oxidative Stress; Analgesia
MeSH Terms: conditions — Agnosia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 3 blood samples before induction, 1 hour after the end of the induction at the time of the blood gas to adapt the ventilation and 24 hours from the start of the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With lidocaine: Patient with injection of a 1.5 mg/kg bolus of lidocaine at induction of anaesthesia
  Interventions: Biological: Blood sample
- Without lidocaine: Patient without injection of a 1.5 mg/kg bolus of lidocaine at induction of anaesthesia
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Blood sample before induction, 1h after induction and 24h after the start of procedure

SUMMARY:
Depending on the anesthesiologist's habits, injection or not of a 1.5 mg/kg bolus of lidocaine at induction of anesthesia followed by a continuous infusion of 1.5 mg/kg/h.

Additional blood sample at 3 different times without additional puncture compared to usual management: 1) during the placement of the venous line before induction (Reactive Oxygen Species), 2) 1h after the end of induction at the time of blood gas to adapt ventilation (Reactive Oxygen Species), 3) at 24h of the beginning of the intervention (Reactive Oxygen Species and antioxidant molecular profile).

DETAILED DESCRIPTION:
Intraoperatively, depending on the habits of the anesthesiologist, lidocaine may be started after induction (bolus of 1.5 mg/kg then relay at 1.5 mg/kg/h until the end of the procedure) or not (control group).

Three blood samples will be taken. The first one (T0) during the placement of the venous line before induction and the second one (T1) one hour after the end of induction when the blood gas on the arterial catheter is taken to adapt the ventilation. These samples will be taken by the nurse in charge of the patient during the procedure. The third sample (T24) will be taken 24 hours after the beginning of the operation, during the blood test (venous or arterial), by the nurse of the department where the patient will be hospitalized. These samples will allow the evaluation of the level of Reactive Oxygen Species (ROS) (T0, T1, T24 - 4ml dry tube) and the antioxidant molecular profile (T24 - same tube as for the evaluation of the ROS (Reactive Oxygen Species) level). The collection of patient data will stop at D1 after the sampling.

The anesthesia protocol will be standardized, in accordance with the department's habits and respecting the recommendations of the French Society of Anaesthesia and Intensive Care (SFAR): patient monitoring (pulse oximeter, invasive arterial catheter, capnograph, curarimeter and sevoflurane concentration monitoring), pre-oxygenation, intravenous induction (propofol, sufentanil, atracurium or rocuronium - dose at the discretion of the anesthesiologist), and maintenance with sevoflurane Intraoperative analgesia will systematically include the injection of sufentanil as well as at the end of the surgery the administration of paracetamol (1g) and nefopam (20 mg) associated or not with an anti-inflammatory. After induction, a dose of 8 mg of dexamethasone will be administered to the patient for the prevention of postoperative nausea and vomiting. In the recovery room, morphine titration can be performed if Visual Analogue Scale (VAS)>3 (3mg/5min). The postoperative analgesia protocol will be left to the discretion of the anesthesiologist.

The parameters collected will be the demographic characteristics (sex, age, weight, height), the terrain (ASA score), the results of the preoperative biological examination (blood ionogram, urea, creatinine, blood count, liver examination), the duration of anesthesia and the doses of drugs received intraoperatively. The parameters measured will be the level of Reactive Oxygen Species in the blood sub populations and the antioxidant molecular profile:

Reactive Oxygen Species :

Analysis will be performed by flow cytometry using DCFDA labeling after erythrocyte lysis. Leukocyte sub populations (lymphocytes, monocytes, polynuclears) will be identified by co-labeling with an anti-Cluster Differentiation 45 antibody (anti-CD45).

Antioxidant molecular profile :

Quantification of the expression of the 26 major antioxidant genes and their isoforms (antioxidogramTM; patent WO2012085188 A1) will be performed on whole blood after RNA extraction, retro transcription into deoxyribonucleic acid (cDNA)

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring urological or ear, nose & throat (ENT) surgery with arterial catheterisation
* ASA 1 to 3
* ≥ 18 years

Exclusion Criteria:

* Heart failure (NYHA ≥ 3)
* Liver failure (aspartate aminotransferase and/or alanine aminotransferase ≥ 2N)
* Chronic renal insufficiency (GFR ≤ 30 ml/min/1.73m2)
* Allergy or intolerance to lidocaine
* Epilepsy
* ASA 4
* Objection to data processing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient requiring urological or ENT surgery with arterial catheterisation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Reactive Oxygen Species | 1 hour after induction
  Analysis will be performed by flow cytometry using DCFDA labelling after erythrocyte lysis. Leukocyte subpopulations (lymphocytes, monocytes, polynuclears) will be identified by co-labelling with an anti-CD45

SECONDARY OUTCOMES:
Reactive Oxygen Species | 24 hours after the start of the procedure
  Analysis will be performed by flow cytometry using DCFDA labelling after erythrocyte lysis. Leukocyte subpopulations (lymphocytes, monocytes, polynuclears) will be identified by co-labelling with an anti-CD45
Molecular antioxidant profile | 24 hours after the start of the procedure
  The quantification of the expression of the 26 main antioxidant genes and their isoforms (antioxydogramTM ; patent WO2012085188 A1) will be performed on whole blood after RNA extraction, retrotranscription in cDNA.

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vignon C, Lachot S, Foucault A, Ravalet N, Gyan E, Picou F, Herault B, Le Nail LR, Bene MC, Herault O. Reactive oxygen species levels differentiate CD34+ human progenitors based on CD38 expression. Cytometry B Clin Cytom. 2020 Nov;98(6):516-521. doi: 10.1002/cyto.b.21948. Epub 2020 Sep 4. PMID 32886395
- [Background] Picou F, Vignon C, Debeissat C, Lachot S, Kosmider O, Gallay N, Foucault A, Estienne MH, Ravalet N, Bene MC, Domenech J, Gyan E, Fontenay M, Herault O. Bone marrow oxidative stress and specific antioxidant signatures in myelodysplastic syndromes. Blood Adv. 2019 Dec 23;3(24):4271-4279. doi: 10.1182/bloodadvances.2019000677. PMID 31869414